CLINICAL TRIAL: NCT05559320
Title: Effects of a Novel, Home-based Training Program Using a Joystick-operated, Modified, Powered Ride-on-car on Bilateral Upper Extremity Function in Children With Hemiplegic Cerebral Palsy
Brief Title: Use of Joystick-operated Ride-on-toys to Improve Affected Arm Use and Function in Children With Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Virginia Tech (National Pediatric Rehabilitation Resource Center i.e. C-PROGRESS) (Unknown); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); American Academy of Cerebral Palsy and Developmental Medicine (Other)
Responsible Party: Principal Investigator, Sudha Srinivasan, Assistant Professor, University of Connecticut
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H22-0059; 1P2CHD101912-01 (NIH)
Record Dates: First submitted 2022-09-16; First posted 2022-09-29 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Hemiplegic Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Joystick Ride-on-car Navigation Training (Experimental): Participants will first participate in a 6-week control phase followed by a 6-week intervention phase. During the intervention phase, they will receive the ride-on-toy navigation training program. The training will be provided by the researchers twice a week, 30-45 minutes/session for 6 weeks. Caregivers will be asked to provide 2 additional sessions/week during the intervention phase. In this study design, the participants will serve as their own controls.
  Interventions: Device: Ride-on-toy navigation training; Behavioral: Upper extremity functional training

INTERVENTIONS:
Device: Ride-on-toy navigation training — The training program will involve a set of activities where children will be encouraged to drive a joystick-operated ride-on-toy to navigate through their physical environment. The training will involve will involve progressively challenging multi-directional navigational games such as shape mazes, treasure hunts, relay races, and obstacle courses that will require children to use their affected arm skillfully to navigate through the courses.
Behavioral: Upper extremity functional training — In addition to the navigation practice, along the multi-directional courses, children will complete tasks at multiple stations that will involve both gross and fine motor activities. The goal of the training will be to use their arm for functional goal-directed tasks and games that will involve elements of reaching, grasping, in-hand manipulation, and release. We will use props such as balls, bean bags, cups, cones, and small toys to practice skills such as catching, throwing, picking up, pushing, pulling, opening, closing, etc.

SUMMARY:
This research is being done to explore if modified, commercially available, joystick-operated, ride-on-cars can be used to promote bilateral arm function in children with hemiplegic Cerebral Palsy (CP). Specifically, the study evaluates the effects of a 6-week, home-based, child-friendly, innovative program that uses modified, commercially available, joystick-operated, powered ride-on-toys to promote spontaneous affected arm use and function in children with hemiplegic CP.

DETAILED DESCRIPTION:
Prior to the start of the study, researchers will conduct a phone screening with the family to confirm their child's eligibility to participate in the study. Once eligibility is confirmed, during the pretest session, standardized assessments will be conducted to evaluate the child's ability to use their affected arm for different functional activities. During this testing visit, researchers will also use small sensors on the child's arms and observe their movements as they complete a reaching task. In addition, caregivers will be asked to complete questionnaires to obtain information on their child's overall health, development, and their ability to use their affected arm for various activities of daily living.

Assessments and questionnaires will be repeated again at the mid-point of the study (that corresponds with completion of the 6-week control phase), and at posttest (that corresponds with completion of the 6-week home-based intervention phase). Researchers will video record all testing and training sessions so that children's performance can be scored later. Children will also be asked to wear wrist monitors on both hands to assess their habitual activity levels on dominant and non-dominant arms for 1 week at the pretest, at the mid-point assessment, during the first and last weeks of the training, and at posttest.

This study consists of 2 phases: the control phase and the intervention phase. During the first 6-week control phase, the researchers will contact families on a weekly basis to obtain information regarding different therapies that their child receives both in and out of school. In the next 6-week intervention phase, researchers will visit the child's home twice a week to provide a training program involving joystick-operated ride-on-toys that will encourage the child to use their affected arm to control and navigate the ride-on-car through their physical environment. During the intervention phase the ride-on-car will be left at the child's home so that children can practice driving the car under caregiver supervision for additional days during the week. All testing sessions will be conducted before and after the control and intervention phases of the study.

ELIGIBILITY:
Inclusion Criteria:

* Are boys or girls between the ages of 3 - 8 years
* Have been diagnosed with hemiplegic Cerebral palsy by a medical doctor with clear asymmetry in upper extremity strength and control, i.e., one upper limb is clearly weaker than the other;
* Have had no physical trauma (including surgery) in the past 6 months;
* Demonstrate awareness of objects in their environment through their visual system;
* Can use their upper extremity or trunk to activate a joystick placed within reachable distance;
* Can maintain a supported sitting position for at least 20 minutes

Exclusion Criteria:

* Have only lower limb involvement
* Are capable of using both hands together very well for functional activities;
* Age >8 years or below 3 years of age
* Exceed safe weight or height limits of the device;
* Have parents who know at the time of the initial contact that they will not be able to complete training and all the posttest sessions

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy Program, Department of Kinesiology, University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amonkar N, Kumavor P, Morgan K, Bubela D, Srinivasan S. Feasibility of Using Joystick-Operated Ride-on-Toys to Promote Upper Extremity Function in Children With Cerebral Palsy: A Pilot Study. Pediatr Phys Ther. 2022 Oct 1;34(4):508-517. doi: 10.1097/PEP.0000000000000944. Epub 2022 Aug 30. PMID 36044637
- [Derived] Shahane V, Kumavor P, Morgan K, Friel KM, Srinivasan SM. A protocol for a single-arm interventional study assessing the effects of a home-based joystick-operated ride-on-toy navigation training programme to improve affected upper extremity function and spontaneous use in children with unilateral cerebral palsy (UCP). BMJ Open. 2023 May 9;13(5):e071742. doi: 10.1136/bmjopen-2023-071742. PMID 37160396
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36044637/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Joystick Ride-on-car Navigation Training
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.92 (2.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Affected Arm Movement Control
Description: The Quality of Upper Extremity Skills Test (QUEST) is a criterion-referenced, valid, and reliable measure for use between 18 months-12 years to assesses quality of UE function in 4 domains: dissociated movement, grasp, protective extension, and weight bearing. The tool includes 36 items that evaluate movement patterns and hand function in children with CP and are scored on a dichotomous scale. Scores for each sub-domain and the total score are calculated as percentages. The total QUEST score was calculated by summing scores for each sub-domain tested divided by the total number of sub-domains tested. The total scores on the QUEST range from 0 to 100. Higher scores represent better quality of movement.
Time Frame: Baseline, at 6-weeks (i.e., at the end of the control phase), at 12-weeks (i.e., at the end of intervention phase)
Measure: Mean (Standard Error); unit: percentage
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 15
percentage
  Baseline | 74.9 (3.1)
  6-weeks (i.e., at the end of the control phase) | 78.3 (3.5)
  12-weeks (i.e., at the end of intervention phase) | 83.8 (2.2)

2. Primary Outcome: Changes in Use of Affected Arm in Functional Activities
Description: The Shriner's Hospital Upper Extremity Evaluation (SHUEE) is a video-based assessment designed to assess spontaneous use and dynamic segmental alignment of the affected UE during functional tasks in children with hemiplegic CP between 3 and 18 years. The SHUEE includes 16 bimanual tasks. Of these 16 tasks, to assess the child's actual function of the affected UE a spontaneous use score is calculated during performance of 9 out of the 16 tasks. This Spontaneous Functional Analysis (SFA) score per task is rated on a scale of 0 to 5, where higher values indicate more spontaneous use of the affected UE. We summed the SFA scores across all 9 tasks, divided this sum by the total possible score, and then multiplied this value by 100 to express SFA as a percentage of normal or optimal score.
Time Frame: Baseline, at 6-weeks (i.e., at the end of the control phase), at 12-weeks (i.e., at the end of intervention phase)
Measure: Mean (Standard Error); unit: percentage of normal or optimal score
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 15
percentage of normal or optimal score
  Baseline | 52.3 (3.4)
  6-weeks (i.e., at the end of the control phase) | 53.3 (3.4)
  12-weeks (i.e., at the end of intervention phase) | 60.7 (3.1)

3. Primary Outcome: Changes in Habitual Arm Activity on the Affected Side
Description: We will provide children with the Actigraph wrist activity monitors that can be worn like a wristwatch. Children will be asked to wear 2 wrist monitors, one each on both wrists, at 6 timepoints: (a) for one week at the pretest, (b) for one week at mid-point assessment, (c) during first week of training, (d) during last week of training, and (e) for one week at posttest. Children will be provided 2 watches during the pretest visit and they will be requested to wear the watches on both wrists for the next 1 week prior to the start of the training program. Children will be asked to wear the monitor continuously when awake and while sleeping for a minimum of 4 days - 1 weekend day and 3 weekdays.
Time Frame: Baseline, at 6-weeks (i.e., at the end of the control phase), at 12-weeks (i.e., at the end of intervention phase)
Measure: Mean (Standard Error); unit: %time Mod-Vig Activity of Affected Side
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 12
%time Mod-Vig Activity of Affected Side
  Baseline | 48.4 (4.3)
  at 6-weeks (i.e., at the end of the control phase) | 50.9 (5.0)
  at 12-weeks (i.e., at the end of intervention phase) | 50.4 (3.5)

4. Primary Outcome: Changes in Kinematic Measures of Movement Control on the Affected Arm
Description: Data will be collected during a unilateral and bilateral reach-grasp task at self-selected speed involving different objects (foam ball, rattle, and square block) placed at half arm's length (near) and at arm's length (far) on the table. Sensors (Inertial Measurement Units (IMUs)) will be placed on both hands, both forearms, both arms, and the C7 spinous process. We will assess range of motion of joints during upper extremity activities.
Time Frame: at 6-weeks (i.e., at the end of the control phase), at 12-weeks (i.e., at the end of intervention phase)
Measure: Mean (Standard Error); unit: degrees
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 8
degrees
  Overhead shoulder ROM at 6-weeks (i.e., at the end of the control phase) | 113.69 (6.53)
  Overhead shoulder ROM at 12-weeks (i.e., at the end of intervention phase) | 123.93 (7.47)
  Elbow ROM at 6-weeks (i.e., at the end of the control phase) | 112.68 (7.53)
  Elbow ROM at 12-weeks (i.e., at the end of intervention phase) | 132.59 (7.08)
  Wrist Sagittal ROM at 6-weeks (i.e., at the end of the control phase) | 58.72 (13.80)
  Wrist Sagittal ROM at 12-weeks (i.e., at the end of intervention phase) | 69.78 (16.59)

5. Primary Outcome: Treatment Satisfaction
Description: Children will complete the valid and reliable 16-item Physical Activity Enjoyment Scale (PAES) to rate their experience with the intervention. The PAES includes a mix of 9 positively phrased (e.g., I enjoy it, It gives me energy, etc.) and 7 negatively phrased (e.g., I feel bored, It's no fun at all, etc.) questions that are rated on a 5-point Likert scale (1: Disagree a lot, 5 - Agree a lot). The negatively coded items were reverse coded and an average total score across all items was calculated. The PAES total score ranges from 1 to 5, with higher scores indicating greater levels of enjoyment with training activities.
Time Frame: At 6-weeks (i.e., at the end of the control phase), at 12 weeks (i.e. following completion of the intervention phase)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 14
score on a scale
  6-weeks (i.e., at the end of the control phase) | 3.7 (0.2)
  12 weeks (i.e. following completion of the intervention phase) | 3.9 (0.1)

6. Primary Outcome: Perceived Satisfaction With Intervention
Description: Children and caregivers will fill out exit questionnaires to assess training satisfaction, enjoyment, repeatability, and caregiver burden.
Time Frame: At 12 weeks (i.e. following completion of the intervention and control phases each lasting for 6 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 15
Participants
  number of children reporting high enjoyment | 12
  number of caregivers agreeing RNT is overall beneficial | 15

7. Primary Outcome: Ease of Implementation of Training
Description: Trainers will fill out posttest exit questionnaires to assess ease of implementation of the training program.
Time Frame: At 12 weeks (i.e. following completion of the intervention and control phases each lasting for 6 weeks)
Population: child and caregiver
Measure: Count of Participants; unit: Participants
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 15
Participants
  number of children wanting to repeat RNT | 14
  number of caregivers reporting some difficulty in independently delivering RNT | 9

8. Primary Outcome: Changes in Treatment Fidelity Across Training Weeks
Description: An unbiased coder randomly coded video data (one each of early, mid, and late sessions) from researcher-delivered sessions within the intervention phase using a fidelity checklist to assess adherence to the training protocol. A 159-item fidelity checklist (total possible score: 159) specific to the training program was used for scoring treatment fidelity. Each item was rated on scale of 0 to 1, where 0 meant that the criterion was not satisfied and 1 meant that the fidelity criterion was satisfied. The total scores on the checklist could range from 0 to 159. We calculated a percent fidelity score by dividing the total score received by the total possible score (i.e., 159) and then multiplied this value by 100.
Time Frame: Early (week 1), Mid (week 3), and late (week 6) training sessions within the 6-week intervention phase
Measure: Mean (Standard Error); unit: percentage of total possible score
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 15
percentage of total possible score
  Early (week 1) | 95.1 (0.7)
  Mid (week 3) | 96.1 (0.4)
  Late (week 6) | 95.6 (0.7)

9. Primary Outcome: Changes in Toy Use (in Minutes/Week) Across Training Weeks
Description: Sensors mounted on the toy will collect data on amount of use (in minutes/week) of the toy during training weeks. We will assess toy use on a weekly basis across the training period.
Time Frame: From start to end of 6-week intervention phase on a weekly basis
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 12
minutes
  Week 1 Duration | 34.3 (3.6)
  Week 2 Duration | 41.5 (5.7)
  Week 3 Duration | 44.2 (5.1)
  Week 4 Duration | 40.4 (4.1)
  Week 5 Duration | 38.5 (5.5)
  Week 6 Duration | 60.4 (9.7)

10. Primary Outcome: # of Training Sessions Completed Assessed Using Training Logs
Description: Researchers will also maintain training logs during the intervention phase to document # of training sessions completed out of the total possible sessions (12).
Time Frame: From start to end of 6-week intervention phase on a weekly basis
Measure: Mean (Standard Error); unit: percentage of sessions attended
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 15
percentage of sessions attended | 98.33 (1.21)

11. Secondary Outcome: Changes in Parent-rated Scores on Functional Use of the Affected Arm
Description: The ABILHAND-Kids is a valid and reliable parent-rated questionnaire assessing parent perceptions of their child's level of ease or difficulty in performing 21 manual activities independently over the last 3 months. The questionnaire has been validated as a measure of manual ability for 6-16-year-old children with CP. The 21 manual activities are rated by parents on a 3-point scale of "impossible" (given a score of 0), "difficult" (given a score of 1), or "easy" (given a score of 2). ABILHAND score is expressed in logits, resulting from the conversion of the ordinal raw score into a linear measure of ability located on a unidimensional scale. The logit is a linear unit that expresses the odds of success of the patient on any given item. This unit is constant throughout the measurement scale. The manual ability scale is, by convention, centered on the average item difficulty (0 logit), the scale ranging from -6.75 to 6.68, with higher scores indicating better manual abilities.
Time Frame: Baseline, at 6-weeks (i.e., at the end of the control phase), at 12-weeks (i.e., at the end of intervention phase)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 15
score on a scale
  Baseline | 0.1 (0.4)
  6-weeks (i.e., at the end of the control phase) | 0.5 (0.3)
  12-weeks (i.e., at the end of intervention phase) | 1.2 (0.3)

12. Secondary Outcome: Changes in Amount of Trainer Assistance Needed During Navigation
Description: Early, mid, & late training sessions will be coded for % duration of assisted (child needs trainer-provided manual assistance) versus independent navigation.
Time Frame: Early (week 1), mid (week 3), and late (week 6) training sessions within the 6-week intervention phase
Measure: Mean (Standard Error); unit: %session spent in independent navigation
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 15
%session spent in independent navigation
  Early (week 1) | 73.4 (4.3)
  Mid (week 3) | 88.7 (3.3)
  Late (week 6) | 95.4 (1.7)

13. Secondary Outcome: Changes in Child Attention During Training Sessions
Description: Training sessions (one early, mid, and late session each) will be video-coded for attention (i.e., % duration of attention to task-relevant targets).
Time Frame: Early (week 1), mid (week 3), and late (week 6) sessions during the 6-week intervention phase
Measure: Mean (Standard Error); unit: % duration of attention to task targets
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 15
% duration of attention to task targets
  Early (week 1) | 80.7 (1.6)
  Mid (week 3) | 83.9 (1.8)
  Late (week 6) | 83.4 (1.4)

14. Secondary Outcome: Changes in Child Affect Across Training Sessions
Description: Training sessions (one early, mid, and late session each) will be video-coded for child affect (i.e., smile rates, % duration of positive/interested and negative affect)
Time Frame: Early (week 1), mid (week 3), and late (week 6) sessions during the 6-week intervention phase
Measure: Mean (Standard Error); unit: % duration in positive/interested affect
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 15
% duration in positive/interested affect
  Early (week 1) | 98.1 (1.1)
  Mid (week 3) | 99.3 (0.4)
  Late (week 6) | 98.9 (0.5)

15. Secondary Outcome: Changes in the Duration of Movement Bouts During Navigation Across Testing Sessions
Description: The path navigation test will be coded for the average duration of child-initiated, movement bouts normalized by driving time (a bout comprises 1 acceleration and 1 deceleration phase).
Time Frame: Baseline, at 6-weeks (i.e., at the end of the control phase), at 12-weeks (i.e., at the end of intervention phase)
Measure: Mean (Standard Error); unit: Bout Rate (bouts/min)
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 15
Bout Rate (bouts/min)
  Baseline | 31.2 (3.7)
  6-weeks (i.e., at the end of the control phase) | 27.7 (4.2)
  12-weeks (i.e., at the end of intervention phase) | 14.8 (3.1)

16. Secondary Outcome: Changes in Rates of Obstacle Contacts Across Testing Sessions
Description: The path navigation test will be coded for the number of times the child bumps/crashes against obstacles during the navigation. We will report on the number of such bumps/crashes per minute of navigation time. Higher values of this variable indicate worse performance (poor navigational control).
Time Frame: Baseline, at 6-weeks (i.e., at the end of the control phase), at 12-weeks (i.e., at the end of intervention phase)
Measure: Mean (Standard Error); unit: bumps/crashes per minute
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 15
bumps/crashes per minute
  Baseline | 1.4 (0.3)
  6-weeks (i.e., at the end of the control phase) | 1.8 (0.3)
  12-weeks (i.e., at the end of intervention phase) | 0.5 (0.1)

17. Secondary Outcome: Changes in Rates of Path Deviations Across Testing Sessions
Description: The path navigation test will involve children navigating through paths that are clearly demarcated using tape/chalk. We counted the number of times per minute that children went outside the demarcated path during the navigation test. Higher values of this variable indicate worse performance (poor navigational control).
Time Frame: Baseline, at 6-weeks (i.e., at the end of the control phase), at 12-weeks (i.e., at the end of intervention phase)
Measure: Mean (Standard Error); unit: path deviations per minute
Arm/Group | Single Joystick Ride-on-car Navigation Training
Number analyzed (Participants) | 15
path deviations per minute
  Baseline | 2.2 (0.2)
  6-weeks (i.e., at the end of the control phase) | 2.0 (0.1)
  12-weeks (i.e., at the end of intervention phase) | 1.2 (0.4)

ADVERSE EVENTS:
Time Frame: 15 weeks
Groups:
- Control Phase (Treatment-as-usual): This is a single arm study design where participants will serve as their own controls. Participants will first be observed during a 6-week control phase where we will only keep track of the usual care they typically receive through school/clinic-based systems. There is no active research-based intervention provided during this phase by the study team.
- Intervention Phase (Treatment-as-usual + Single Joystick Ride-on-toy Navigation Training): During the following 6-week intervention phase, children will receive the ride-on-toy navigation training program delivered by the study team. The training will be provided by the researchers twice a week, 30-45 minutes/session for 6 weeks. Caregivers will be asked to provide 2 additional sessions/week during the intervention phase.
Arm/Group | Control Phase (Treatment-as-usual) | Intervention Phase (Treatment-as-usual + Single Joystick Ride-on-toy Navigation Training)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-03-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT05559320/Prot_SAP_ICF_001.pdf